CLINICAL TRIAL: NCT04599140
Title: Phase Ib/II Trial of SX-682 in Combination With Nivolumab for Refractory RAS Mutated (RAS) Microsatellite Stable (MSS) Metastatic Colorectal Cancer (mCRC) (STOPTRAFFIC-1)
Brief Title: SX-682 and Nivolumab for the Treatment of RAS-Mutated, MSS Unresectable or Metastatic Colorectal Cancer, the STOPTRAFFIC-1 Trial
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry); Syntrix Biosystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1151; NCI-2020-07989 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1151 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-10-09; First posted 2020-10-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Colon Adenocarcinoma; Metastatic Colorectal Carcinoma; Metastatic Rectal Adenocarcinoma; Stage III Colon Cancer AJCC v8; Stage III Rectal Cancer AJCC v8; Stage IIIA Colon Cancer AJCC v8; Stage IIIA Rectal Cancer AJCC v8; Stage IIIB Colon Cancer AJCC v8; Stage IIIB Rectal Cancer AJCC v8; Stage IIIC Colon Cancer AJCC v8; Stage IIIC Rectal Cancer AJCC v8; Stage IV Colon Cancer AJCC v8; Stage IV Rectal Cancer AJCC v8; Stage IVA Colon Cancer AJCC v8; Stage IVA Rectal Cancer AJCC v8; Stage IVB Colon Cancer AJCC v8; Stage IVB Rectal Cancer AJCC v8; Stage IVC Colon Cancer AJCC v8; Stage IVC Rectal Cancer AJCC v8; Unresectable Colon Adenocarcinoma; Unresectable Rectal Adenocarcinoma
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Rectal Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (SX-682, nivolumab) (Experimental): MONOTHERAPY STAGE: Patients receive SX-682 orally PO BID on days 1-21 in the absence of disease progression or unacceptable toxicity.
  COMBINATION STAGE: Patients receive SX-682 PO BID on days 1-56 and nivolumab IV over 30 minutes on days 1 and 29. Treatment repeat every 56 days weeks for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: CXCR1/2 Inhibitor SX-682; Biological: Nivolumab

INTERVENTIONS:
Drug: CXCR1/2 Inhibitor SX-682 — Given PO
  Other Names: SX 682; SX-682; SX682
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase Ib/II trial studies the side effects and best dose of SX-682 that can be given alone and in combination with nivolumab in treating patients with RAS-Mutated, microsatellite stable (MSS) colorectal cancer that has spread to other places in the body (metastatic) or cannot be removed by surgery (unresectable). SX-682 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving SX-682 alone and together with nivolumab may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety profile of CXCR1/2 Inhibitor SX-682 (SX-682) alone and in combination with nivolumab in subjects with refractory RAS mutated microsatellite stable (MSS) metastatic colorectal cancer (mCRC), including the maximum dose that can be administered until adverse effects prevent further dose increases (i.e., the maximum tolerated dose [MTD] or recommended phase 2 dose), and the dose-limiting toxicity (DLT).

SECONDARY OBJECTIVES:

I. Evaluate the efficacy of SX-682 in combination with nivolumab on the basis of the objective response rate (ORR), the duration of response, and the rate of progression.

II. Characterize the single-dose and multidose pharmacokinetic (PK) profile of SX-682.

EXPLORATORY OBJECTIVES:

I. Assess overall survival (OS). II. Explore potential biomarkers associated with pharmacodynamic and clinical response to SX-682 alone and combined with nivolumab, where the biomarker measures include, but are not limited to, tumor CMS4, gene expression, deoxyribonucleic acid (DNA) mutations (KRAS, NRAS and BRAF mutation status via ribonucleic acid [RNA] and DNA sequencing), IRF2 (interferon regulatory factor 2) expression, lymphocyte clonality (via sequencing), myeloid-derived suppressor cell (MDSCs), regulatory T-cells (Tregs) and CD69/CD8 T cells, and in the circulation, circulating tumor DNA (ctDNA), T- and B-cell subpopulations, neutrophils, the neutrophil-to-lymphocyte ratio (NLR), MDSCs, Tregs, the CD4:CD8 ratio, chemokines and cytokines.

OUTLINE: This is a phase I, dose-escalation study of CXCR1/2 Inhibitor SX-682, followed by a phase II study.

MONOTHERAPY STAGE: Patients receive SX-682 orally (PO) twice daily (BID) on days 1-21 in the absence of disease progression or unacceptable toxicity.

COMBINATION STAGE: Patients receive SX-682 PO BID on days 1-56 and nivolumab intravenously (IV) over 30 minutes on days 1 and 29. Treatment repeat every 56 days weeks for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study, patients with no have tumor response are followed up every 3 weeks for 90 days, and patients with tumor response every 3 months for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent and HIPAA Authorization

   1. Subjects must have the nature of the study explained to them.
   2. Non-English speaking patients will be eligible for participation with involvement of the MD Anderson Language Assistance department in the informed consent process (per MD Anderson SOP 04_Informed Consent Process).
   3. Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, pharmacokinetic collections, and other requirements of the study.
   4. Subjects must provide a signed and dated IRB approved written informed consent form (ICF) in accordance with regulatory and institutional guidelines for both the study and exploratory biomarker analyses (e.g., CMS4 and others) on archival tissue.
   5. Subjects must provide a signed and dated Health Insurance Portability and Accountability Act (HIPAA) authorization.
   6. The ICF and HIPAA authorization must be obtained before conducting any procedures that do not form a part of the subject's normal care.
   7. After signing the ICF and HIPAA Authorization, subjects will be evaluated for study eligibility during the Screening Period (no more than 28 days before study drug administration) according to the following further inclusion/exclusion criteria:
2. Target Population

   1. Men and women, ages > 18 years of age. Both men and women of all races and ethnic groups, regardless of preferred language, are eligible for this trial.
   2. Histologically or cytologically confirmed adenocarcinoma of the colon or the rectum that is metastatic or unresectable.
   3. Tumor is determined to be RAS-mutated (KRAS or NRAS) and microsatellite stable/proficient in mismatch repair, as assessed by IHC and/or PCR/NGS in a CLIA environment.
   4. Received at least two prior regimens of therapy for unresectable or metastatic CRC including fluoropyrimidine-, oxaliplatin-, and irinotecan-based regimens. Patients who relapse within 6 months of adjuvant chemotherapy composed of oxaliplatin and a fluoropyrimidine will have their adjuvant therapy count as one prior regimen.
   5. For the expansion cohort, pre-treatment primary tumor tissue (i.e., archived paraffin-embedded) or from an unresectable metastatic site must be available for biomarker analyses. Biopsy should be excisional or core needle. Fine needle aspirates or other cytology samples are insufficient.
   6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1 (Appendix 1).
   7. Must have measurable disease with at least 1 unidimensional measurable lesion per RECIST v1.1 (see Appendix 2).
   8. Prior radiotherapy must have been completed at least 2 weeks prior to study drug administration.
   9. Screening laboratory values must meet the following criteria and should be obtained within 14 days prior to first dose:

      WBC > 3000/µL Neutrophils > 1500/ µL Platelets > 100,000/µL Hemoglobin > 9.0 g/dL (may have been transfused) Creatinine < 1.5 mg/dL AST/ALT < 2.5 X ULN for subject with no liver metastases < 5 X ULN for subjects with liver metastases Bilirubin < 1.5 mg/dL (unless diagnosed with Gilbert's syndrome, who can have total bilirubin < 3.0 mg/dL) INR or PT < 1.5 X ULN unless the subject is receiving anticoagulant therapy aPTT or PTT < 1.5 X ULN unless the subject is receiving anticoagulant therapy
   10. Glomerular filtration rate (GFR) calculated by Cockcroft-Gault formula >60 ml/min.
   11. Life expectancy > 12 weeks as judged by the treating physician.
   12. Subject Re-enrollment: This study permits the re-enrollment of a subject that has discontinued the study as a pre-treatment failure (i.e., subject has not been treated with SX-682). If re-enrolled, the subject must be re-consented.

Exclusion Criteria

1. Target Disease Exceptions

   a) Active brain metastases or leptomeningeal metastases. Subjects with brain metastases are eligible if these have been treated and there is no magnetic resonance imaging (MRI - except where contraindicated, in which CT scan is acceptable) evidence of progression for at least 8 weeks after treatment is complete and within 28 days prior to first dose of study drug administration. An MRI is not required to rule out brain metastases or leptomeningeal metastases. There must also be no requirement for high doses of systemic corticosteroids that could result in immunosuppression (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration.

   b) Patients with bulky liver metastases (liver metastases >3cm) are not eligible.
2. Medical History and Concurrent Diseases

   a) Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results. Specifically:

   a. Subjects with active, non-infectious pneumonitis. b. Subjects with interstitial lung disease or a history of pneumonitis that required oral or intravenous glucocorticoids to assist with management.

   c. Subjects with clinically significant heart disease that affects normal activities. Clinically significant cardiovascular/ cerebrovascular disease as follows: cerebral vascular accident / stroke / carotid artery disease / transient ischemic attack (<6 months prior to enrollment), myocardial infarction (<6 months prior to enrollment), unstable angina, congestive heart failure (New York Heart Association Classification Class >II) or serious cardiac arrhythmia.

   b) Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.

   c) Subjects with active, known or suspected autoimmune disease (Appendix 3). Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.

   d) Subjects with a condition (including organ or bone marrow transplant) requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.

   e) Use of other investigational drugs (drugs not marketed for any indication) or medications at immunosuppressive doses within 28 days before study drug administration.

   f) Prior exposure to any immune checkpoint blockade agent or any other immunomodulatory agent used for antineoplastic therapy for mCRC.

   g) Anticancer treatment within 21 days before the start of trial treatment [e.g., cytoreductive therapy, radiotherapy (with the exception of palliative radiotherapy delivered in a normal organ-sparing technique), immune therapy, or cytokine therapy]. Note: Patients on maintenance anti-hormonal treatment to prevent recurrence and secondary cancers are eligible for participation.

   h) Major surgery as determined by the investigator within 28 days before the start of trial treatment (prior diagnostic biopsy is permitted).

   i) Subjects who have received a live-virus vaccine within 30 days before study drug administration.

   j) Treatment with botanical preparations (e.g., herbal supplements or traditional Chinese medicines) intended for general health support or to treat the disease under study within 2 weeks prior to randomization/treatment.

   k) Patients who are taking any drug that is known to prolong QTc interval within at least 2 weeks before the start of trial drug and during the conduct of the trial.

   l) Individuals lacking the ability, based on reasonable medical judgment, to understand and appreciate the nature and consequences of participation in this study will not be eligible for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 2 years
  For each system organ class and preferred term, summaries will be made with respect to the number and proportion of subjects having at least 1 occurrence of an adverse event during the study. The incidence of AEs will be presented overall, by system organ class and preferred term, intensity (based on National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0), immune-related adverse events, treatment-emergent adverse events, and additional grouping by severity and relationship to study drug. Individual listings of adverse events will be provided. Dose limiting toxicities and study drug-related grade >= 2 adverse events will be listed individually.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years
  Patient response will be determined using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Unconfirmed responses will not be used in the final analysis. ORR is defined by the number of (partial response + complete response)/ (total number of treated patients) in the cohort. Will estimate the response rate along with the two-sided exact 95% confidence interval.
Progression-free survival (PFS) | Up to 104 weeks
  Assessed according to RECIST 1.1. Median PFS and 95% confidence intervals will be estimated using the Kaplan-Meier method.
Overall survival (OS) | Up to 104 weeks
  OS time will be presented using the Kaplan-Meier method. Median OS with 95% confidence interval will be estimated using the Kaplan-Meier method.

OTHER OUTCOMES:
Biomarker analysis | Up to 2 years
  Summary statistics will be tabulated for CMS4, interferon regulatory factor 2 expression, lymphocyte clonality (via sequencing), myeloid-derived suppressor cells , regulatory T-cells and CD69/CD8 T cells, and in the circulation, circulating tumor deoxyribonucleic acid T- and B-cell subpopulations, neutrophils, the neutrophil-to-lymphocyte ratio, the CD4:CD8 ratio, KRAS, NRAS and BRAF status. Paired t-test or Wilcoxon signed rank test will be used to assess the changes in biomarkers pre and post-treatment. The differences in biomarker levels between responders and non-responders will be assessed using X2 or Fisher's exact test as appropriate. The correlation between biomarker mutation statuses will be assessed using Paired t-test or Wilcoxon signed rank test. Differences in biomarker levels will be assessed using X2 or Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Alisha Bent, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org